CLINICAL TRIAL: NCT03839875
Title: A National, Multi-central, Open-label, Single-arm, Phase IV Study to Evaluate Efficacy and Safety of Gynomax® XL Ovule in the Treatment of Trichomonal Vaginitis, Bacterial Vaginosis, Candidal Vulvovaginitis and Mixed Vaginal Infections
Brief Title: Evaluation of Efficacy and Safety of Gynomax® XL Ovule
Acronym: Gyno-Türk
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Exeltis Turkey (Industry)
Collaborators: Monitor CRO (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MON564.130.1
Record Dates: First submitted 2019-02-11; First posted 2019-02-15 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Trichomonal Vaginitis; Bacterial Vaginosis; Candidal Vulvovaginitis; Mixed Vaginal Infections
MeSH Terms: conditions — Trichomonas Vaginitis; Vaginosis, Bacterial; Candidiasis, Vulvovaginal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Treatment (Experimental)
  Interventions: Drug: Gynomax® XL Vaginal Ovule

INTERVENTIONS:
Drug: Gynomax® XL Vaginal Ovule — tioconazole, tinidazole, lidocaine

SUMMARY:
Efficacy and safety of Gynomax® XL ovule in the treatment of trichomonal vaginitis, bacterial vaginosis, candidal vulvovaginitis and mixed vaginal infections will be evaluated in this open label, single-arm, multicentral study.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with age ≥ 18 and ≤ 45 years
* Patients requiring treatment for bacterial vaginosis, candidal vulvovaginitis or mixed infections according to the investigator's decision
* Signed informed consent

Exclusion Criteria:

* Known hypersensitivity to active ingredients of the study medications
* Vaginismus, endometriosis, dyspareunia
* Detection of urinary tract infection in urinalysis
* Acute or chronic infections such as pancreatitis, hypertriglyceridemia, liver diseases, benign or malign tumors
* Usage of herbal medicines that interfere with microsomal enzymes, especially cytochrome P450 (phenytoin, phenobarbital, primidone, carbamazepine, rifampicin, topiramate, felbamate, griseofulvin, HIV protease inhibitors such as ritonavir, nucleoside reverse transcriptase inhibitors such as efavirenz)
* History of cardiovascular event
* Advanced hypertension and diabetes
* Presence or known risk or of venous or arterial thromboembolism
* Undiagnosed abnormal vaginal bleeding, bleeding disorders, genital tumors
* Use of drugs containing ombitasvir / paritaprevir / ritonavir or dasabuvir during or two weeks before initiation of the study
* Pregnancy and/or breastfeeding
* Participation in any other trial 30 days before initiation of the study
* Postmenopausal women
* Abuse of alcohol
* Usage of medications containing acenocoumarol, anisindione, dicoumarol, phenindione, phenprocoumon, warfarin, cholestyramine, cimetidine, cyclosporine, disulfiram, fluorouracil, fosphenitoin, ketoconazole, lithium, rifampin, tacrolimus or propranolol
* Presence of a sexually transmitted disease such as syphilis, gonorrhea, etc. according to the investigators decision

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2019-04-03 (Actual); Primary Completion 2019-08-09 (Actual); Study Completion 2019-08-09 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with complete response to treatment | 10 Days after completion of treatment

SECONDARY OUTCOMES:
Percentage of patients with partial response to treatment | 10 Days after completion of treatment
Percentage of patients with no response to treatment | 10 Days after completion of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Ege University Family Planning and Infertility Application and Research Centeraştırma Merkezi, Izmir, Turkey (Türkiye)